CLINICAL TRIAL: NCT03820622
Title: Comparison of the Safety and Efficacy Between Paclitaxel-Eluting Coronary Balloon Dilation Catheter (DIOR) and Paclitaxel-Eluting Balloon (Bingo) in Coronary Bifurcation Lesions: A Prospective, Multicenter, Randomized, Controlled Trial (BEYOND II)
Brief Title: The Safety and Efficacy of DIOR Balloon in Coronary Bifurcation Lesions
Acronym: BEYOND-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CCRF Inc., Beijing, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIOR 2nd -1706
Record Dates: First submitted 2019-01-24; First posted 2019-01-29 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Percutaneous Coronary Intervention
Keywords: coronary artery stenosis; drug eluting balloon; bifurcation
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIOR group (Experimental): in this group, patients will be treated with Paclitaxel-Eluting Coronary Balloon Dilation Catheter (DIOR)
  Interventions: Device: Paclitaxel-Eluting Coronary Balloon Dilation Catheter (DIOR)
- Bingo group (Active Comparator): in this group, patients will be treated with Paclitaxel-Eluting Balloon (Bingo)
  Interventions: Device: Paclitaxel-Eluting Balloon (Bingo)

INTERVENTIONS:
Device: Paclitaxel-Eluting Coronary Balloon Dilation Catheter (DIOR) — patients in the study group will be treated by the Paclitaxel-Eluting Coronary Balloon Dilation Catheter (DIOR)
  Arms: DIOR group
Device: Paclitaxel-Eluting Balloon (Bingo) — patients in the study group will be treated by the Paclitaxel-Eluting Balloon (Bingo)
  Arms: Bingo group

SUMMARY:
To evaluate the safety and effectiveness of paclitaxel-eluting coronary artery balloon dilation catheter (DIOR) in revascularization of coronary bifurcation lesions compared with paclitaxel-eluting balloon (Bingo), and to provide the clinical data for the formal application in China and for the approvement of China marketing.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomize, control and non-inferior study. 220 patients with bifurcation lesions will be randomized 1:1 to each group. after the main branch has been treated successfully, and if the side branch's stenosis is more than 70% and can be pre-dilated by POBA (plain old balloon angioplasty) successfully, then randomizing. the patients in the study group will be treated with paclitaxel-eluting coronary artery balloon dilatation catheter (DIOR), while those in the control group will be treated with paclitaxel-eluting balloon (Bingo). Clinical follow-up will be conducted at baseline, operation, hospital discharge, 1 month, 6 months, 9 months and 12 months after operation, and angiographic follow-up will be conducted at 9 months. The primary endpoint is late lumen loss (LLL) in the balloon dilatation coverage area of side branch of at 9 month after operation. The secondary endpoints include device success, clinical success, target lesion failure (TLF), target lesion revascularization (TLR), clinical composite endpoints and imaging endpoints. The information of adverse events, serious adverse events and device defects will be collected during the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects that participate in this study must fulfill all the following criteria:

General inclusion criteria:

1. Age from 18 to 80 years old, man or non-pregnant woman;
2. Subjects with stable or unstable angina, old myocardial infarction, or asymptomatic ischemic evidence with clinical diagnosis;
3. Subjects without contraindications of coronary artery bypass grafting (CABG);
4. Subjects must agree to the follow up of angiographic and clinical required in the study;
5. Subjects are able to understand the purpose of this study, provide an informed consent to show recognize to the study protocol.

Angiographic inclusion criteria:

1. One or two bifurcation lesions, locate in different epicardial vessels, the bifurcation lesion in each epicardial vessel can not over 1; or 1 de nove coronary artery bifurcation can be included after 1 lesion of non-target vessel has been successfully treated by PCI (Percutaneous Coronary Intervention);
2. Residual diameter stenosis in main branch (MB) ≥ 70% (visually), or ≥ 50% simultaneously with clinical symptom, and the diameter stenosis in side branch (SB) ≥ 50% (visually); and the main branch's residual stenosis ≤ 20% with TIMI 3 flow post the stent placement, while the side branch diameter stenosis ≥ 70% post the MB stenting;
3. Fulfill the definition of truly bifurcation lesions by Medina type (1.1.1、1.0.1、0.1.1);
4. Diameter in side branch between ≥ 2.5 mm to ≤ 4.00 mm (visually) and lesion length ≤ 26 mm (visually);
5. Each side branch of the bifurcation lesion can be treated by only 1 study drug coated balloon (DCB) or control DCB, and the lesion shall be fully covered by the DCB ( the distal end of the balloon shall exceed the lesion at least 1 mm).

Exclusion Criteria:

If subjects fulfill any of below criteria, this subject shall be exclude from this study.

General exclusion criteria:

1. Pregnant or lactating women
2. Any newly myocardial infarction onset within 1 week or, the myocardial enzyme of CK (Creatine Kinase) or CK-MB does not return to normal level after any myocardial infarction;
3. Cardiogenic shock;
4. Severe chronic heart failure, NYHA (New York Heart Association) ≥ grade III, or left ventricular ejection fraction < 35% (accessed by echocardiography or left ventricular angiography)
5. Patients with renal insufficiency (estimated glomerular filtration rate < 30ml/min/1.73m2 calculated by MRDR (Modification of Diet in Renal Disease) formula or subject is receiving renal dialysis)
6. Having a history of hemorrhagic diseases such as cerebral hemorrhage, gastrointestinal hemorrhage; stroke occurring or any situation occurring that may lead to prolongation of anticoagulation therapy within 6 months before operation;
7. History of coronary or peripheral vascular interventional therapy within 12 months before hospitalized.
8. Patients are allergic or contraindicate to contrast agent, paclitaxel, heparin, antiplatelet and anticoagulant drug;
9. The Subjects have other serious diseases and the expected survival is less than 12 months;
10. Investigators determine the subjects' compliance is poor, cannot complete the study as required;

Angiographic exclusion criteria

1. Main branch lesion or non-target lesion(s) located in left main;
2. Main branch lesion or non-target lesion(s) is triple vessel lesion, all need to be treated;
3. Side branch lesion is triple bifurcation or multiple bifurcation;
4. Main branch lesion located within 3 mm of the origin of the LAD (Left Anterior Descending), LCX (Left Circumflex Branch) or RCA (Right Coronary Arter);
5. Side branch target lesion is diffusion lesion and length > 26mm; or a ≥90% stenosis lesion is found near the SB lesion within 5 mm;
6. Side branch as the target vessel has received any interventional treatment;
7. Side branch as the target lesion or target vessel involve in aneurysm;
8. The lesion in side branch or main branch is total occlusive lesions, with TIMI blood flow of grade 0;
9. Side branch target lesion is moderate or heavy calcified or target vessel excessive tortuosity, which is unfavorable for interventional treatment anatomically;
10. Subject's blood pressure is too low to be injected with nitroglycerin ≥ 100 ug, this subject can not be included in the study;
11. Side branch target lesion can not reach the following outcomes, after the completely balloon pre-dilatation:

1) Residual stenosis (DS %) is ≤50% (visually); 2) TIMI Grade-3 flow ((visually); 3) No angiographic complications (e.g., no-reflow, distal embolization, side branch closure) 4) No dissections NHLBI grade C-F;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
late lumen loss | 9 months after operation
  in balloon dilated coverage area of the side branch lesion measured by QCA (Quantitative Coronary Angiography)

SECONDARY OUTCOMES:
device success | immediately post procedure
  define as dilation success in the side branch lesion by study balloon or control ballon, that is the residual stenosis ≤50%，TIMI (Thrombolysis In Myocardial Infarction) 3 flow and without type C or above dissection
clinical success | 1 month after operation
  define as absence of patients oriented composite endpoints (PoCE) during hospitalization, based on the device success.
device oriented composite endpoints (DoCE) | 1, 6, 9, 12 month after operation
  that is TLF, define as the composite endpoint include cardiac death, target vessel myocardial infarction and ischemic driven target lesion revascularization (ID-TLR)
patients oriented composite endpoints (PoCE) | 1, 6, 9, 12 month after operation
  define as a composite endpoints of all cause death, any myocardial infarction and any revascularization
all cause death | 1, 6, 9, 12 month after operation
  include cardiac death, vascular death, noncardiovascular death
myocardial infarction (MI) | 1, 6, 9, 12 month after operation
  target vessel MI, non-target vessel MI
target lesion revasculation | 1, 6, 9, 12 month after operation
  ischemic driven, non-ischemic driven
target vessel revasculation | 1, 6, 9, 12 month after operation
  ischemic driven, non-ischemic driven
any coronary revasculation | 1, 6, 9, 12 month after operation
thrombosis in the side branch lesion | 1, 6, 9, 12 month after operation

OTHER OUTCOMES:
angiographic endpoints-late loss of side branch | 9 months after operation
  assess in millimeter
angiographic endpoints-minimal lumen diameter (MLD) of side branch | 9 months after operation
  assess in millimeter
angiographic endpoints-diameter stenosis (DS) | 9 months after operation
  assess in percentage
angiographic endpoints-angiographic binary restenosis (ABR) | 9 months after operation
  assess in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, professor, Principal Investigator — The General Hospital of Northern Theater Command
Locations (13):
- China (13):
  - Daqing Oil General Hospital, Daqing, Heilongjiang
  - Wuhan Asian Heart Hospital, Wuhan, Hubei
  - Nanjing First Hospital, Nanjing, Jiangsu
  - First Bethune Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian University, Dalian, Liaoning
  - General Hospital of Northern Theater Command, Shengyang, Liaoning
  - The First Hospital of China Medical University, Shengyang, Liaoning
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Anzhen Hospital Capital Medical University, Beijing
  - Shanghai East Hospital,, Shanghai
  - Tianjin Chest Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided